CLINICAL TRIAL: NCT06182371
Title: Effectiveness of Detachment of the Breathing Circuit on the Rate of the Double-lumen Endotracheal Tube Malposition After the Change of Position in Patients Undergoing Thoracic Surgery: a Randomized Controlled Trial
Brief Title: Effectiveness of Detachment of the Breathing Circuit on the Rate of DLT Malposition After Postural Change
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Meng Lv, Deputy Chief Physician, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MLv
Record Dates: First submitted 2023-11-21; First posted 2023-12-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Intratracheal Intubation; Patient Positioning
Keywords: Double-Lumen Endobronchial Tube; Positional changes; Disengage; Breathing circuit; Malposition

STUDY DESIGN:
Intervention Model Description: Intervention: After the insertion of a DLT under general anesthesia, the anesthesiologist disengaged the breathing circuit when the patient transitioned from the supine to the lateral position.
Who Masked: Participant
Masking Description: As this research uses a behavioral intervention, it will conceal the grouping from the subjects. Random numbers will be placed in opaque envelopes by independent persons not involved in this experiment to achieve allocation concealment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disengagement of the breathing circuit (Experimental): When the patient's position is changed from the supine position to the lateral decubitus position, the anesthesiologist disengages the breathing circuit.
  Interventions: Behavioral: Disengage the breathing circuit
- Connect the breathing circuit (No Intervention): When the patient's position is changed from the supine position to the lateral decubitus position, the anesthesiologist maintains the normal connection of the breathing line.

INTERVENTIONS:
Behavioral: Disengage the breathing circuit — Disengage the breathing circuit when the position of the patient undergoing thoracic surgery changes
  Arms: Disengagement of the breathing circuit

SUMMARY:
The goal of this clinical trial is to assess the incidence of double-lumen endobronchial tube displacement in patients undergoing thoracic surgery with a change in position, compared with double-lumen endobronchial tube malposition in chest surgery patients with a fixed breathing circuit. The study is to investigate: whether detaching the breathing circuit in patients undergoing thoracic surgery would reduce the rate of double-lumen endobronchial tube malposition, the incidence of postoperative pulmonary complications, and improve patient outcomes.

Participants will be randomly divided into a disconnected breathing circuit group and a breathing circuit connected group and after entering the operating room, the intravenous access will be opened, and blood pressure, heart rate, electrocardiogram, oxygen saturation, arterial pressure, and end-expiratory carbon dioxide will be monitored. Anesthesia induction will be performed by an anesthesiologist, and then the double-lumen endobronchial tube will be inserted under laryngoscopic guidance. Will the catheter be delivered to the expected depth, the double-lumen endobronchial tube will be connected to the anesthesia machine for mechanical ventilation.

Researchers will compare the malposition rate of the double-lumen endobronchial tube when the patient transitions from the supine to lateral decubitus position, the effect of single-lung ventilation, oxygen saturation at 5 and 10 minutes after single-lung ventilation, and postoperative recovery time.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II elective surgery for patients
* Patients undergoing thoracic surgery requiring a left-sided double-lumen endobronchial tube;
* Sign the informed consent form for this clinical study.

Exclusion Criteria:

* Mouth opening <3cm;
* History of previous difficult intubation;
* Patients with diseases of the upper respiratory tract and main bronchi;
* Cardiac insufficiency;
* People with liver dysfunction;
* Renal insufficiency;
* Previous stroke;
* Patients with severe obstructive ventilation dysfunction;
* Bronchial asthma or airway hyperresponsiveness;
* Patients who have participated in other clinical studies in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Malposition rate of a double-lumen endobronchial tube | Immediately after a change in body position
  Double-lumen endobronchial tube malposition is more than 5 mm away from the optimal position of the catheter. Severe malposition is the inability to see the upper left or lower left bronchial opening in the left common bronchi: the right upper lobe bronchial opening cannot be seen clearly in the right common bronchi; or bronchial cuffs more than 50% in the trachea.

SECONDARY OUTCOMES:
Effects of lung collapse | 5 and 10 minutes after the pleura opens
  If the lung on the operative side is completely atrophied and the surgical field is satisfied, it indicates that the degree of lung atrophy is good. The surgeon will score the quality of lung collapse using a four-point ordinal scale (1= extremelypoor-no collapse of lung; 2= poor-partial collapse of lung with interference with surgical exposure; 3= good-total collapse, but the lung still had some residual air; and 4= excellent-complete collapse of lung with perfect surgical exposure).
Blood oxygen saturation | 1 minute and 5 minutes after the change of position；1 minute, 5 minutes and 10 minutes after single-lung ventilation
  An oxygen saturation below 94% is considered oxygen insufficiency
PACU length of stay | The time from the transfer to the PACU to the transfer out to ward, an average of an hour
  The patient is awake and conscious

OTHER OUTCOMES:
Partial pressure of carbon dioxide at the end of expiration | 1 minute and 5 minutes after the change of position；1 minute, 5 minutes and 10 minutes after single-lung ventilation
  Determine the status of blood-lung ventilation and pulmonary blood flow
Blood pressure | 1 minute and 5 minutes after the change of position；1 minute, 5 minutes and 10 minutes after single-lung ventilation
  Make sure the patient's blood pressure is within the normal range
Heart rate | 1 minute and 5 minutes after the change of position；1 minute, 5 minutes and 10 minutes after single-lung ventilation
  Make sure the patient's heart rate is within the normal range

CONTACTS AND LOCATIONS:
Overall Officials: Jin Bao Mao, Ph.D., Principal Investigator — Shandong Provincial Hospital